CLINICAL TRIAL: NCT04757727
Title: Gynecological Follow-up of Patients With Dystrophic Epidermolysis Bullosa (EBD)
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21dermato01
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Dystrophic Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EDB: Adult women (> 18 years old) with hereditary dystrophic epidermolysis bullosa (dominant or recessive) followed at the Nice University Hospital or at the St Louis Hospital of the APHP
  Interventions: Other: Decriptive study of EDB

INTERVENTIONS:
Other: Decriptive study of EDB — data on EDB will be register

SUMMARY:
Dystrophic epidermolysis bullosa is a rare genetic pathology resulting in fragility of the skin and mucous membranes, causing bubbles and wounds following trauma. Scarring is pathological with a tendency to retraction. The gynecological and in particular the vulvovaginal mucous membranes can be affected but no description of any series is available in the literature. Likewise, some of these patients have a sexual and obstetrical life, despite sometimes-severe damage, but again no specific data is available. The investitigator thus wish to carry out a non-interventional multicenter prospective descriptive study. Better knowledge of gynecological semiology in patients with EBD will allow better adaptation of gynecological follow-up, screening for STDs and gynecological cancers, as well as possible specific complications. This study would eventually allow the draw up of recommendations for our gynecologist / obstetrician colleagues.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* with hereditary dystrophic epidermolysis bullosa (dominant or recessive)
* followed at the Nice University Hospital or at the St Louis Hospital of the APHP.
* not opposed to participation after being informed of the study

Exclusion Criteria:

* men
* age < 18years old

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult women (> 18 years old) with hereditary dystrophic epidermolysis bullosa (dominant or recessive) followed at the Nice University Hospital or at the St Louis Hospital of the APHP.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Descriptve evaluation of the recruited population | 12 months
  Adult women (> 18 years old) with hereditary dystrophic epidermolysis bullosa (dominant or recessive) followed at the Nice University Hospital or at the St Louis Hospital of the APHP.
  Descriptve evaluation of the recruited population Description of the anatomical and gynecological functional impairment of adult women with dystrophic epidermolysis bullosa.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de NICE, Nice
  - Hôpital Saint Louis, Paris

IPD SHARING:
Plan to Share IPD: No
no data sharing plan is schedule